CLINICAL TRIAL: NCT03339115
Title: European Feasibility Study of High Surgical Risk Patients With Severe Mitral Regurgitation Treated With the Cardiovalve Transfemoral Mitral Valve System (AHEAD Study)
Brief Title: AHEAD: European Feasibility Study of the Cardiovalve Transfemoral Mitral Valve System
Acronym: AHEAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiovalve Ltd. (Industry)
Collaborators: Meditrial Europe Ltd. (Industry); Meditrial SrL (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP 17-02
Record Dates: First submitted 2017-11-07; First posted 2017-11-13 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Mitral Regurgitation; Mitral Valve Disease
Keywords: Mitral Insufficiency; Heart Failure; Mitral Valve; Heart Diseases; Valvular Heart Disease
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Failure; Heart Diseases; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cardiovalve Transfemoral Mitral Valve (Experimental): Mitral replacement valve delivered through a transfemoral access and transseptal approach
  Interventions: Device: Cardiovalve Transfemoral Mitral Valve

INTERVENTIONS:
Device: Cardiovalve Transfemoral Mitral Valve — The Cardiovalve Transfemoral Mitral Valve System is intended for use symptomatic patients with severe mitral regurgitation who are at elevated risk for surgical mitral valve repair or replacement and who are anatomically eligible for transfemoral mitral valve replacement with transseptal access to the left atrium.

SUMMARY:
This study will evaluate the safety of the Cardiovalve Transfemoral Mitral Valve System with its associated procedure, and observe the device performance in reducing mitral regurgitation. Data collected in this clinical study will include 30-day safety and performance, and long-term clinical outcomes over a follow-up of 2 years.

DETAILED DESCRIPTION:
The Cardiovalve offers a mitral replacement valve delivered through a transfemoral access and transseptal approach, and is intended to reduce mortality and adverse event rates in selected patients for whom surgical options are not feasible.

Innovation: A truly trans femoral, trans venous delivery of the prosthetic mitral valve which minimizes procedural risk. The Cardiovalve Implant features a dual nitinol frame for robust radial strength with decoupling of the atrial flange and ventricular portion which contains 24 grasping legs designed for atraumatic anchoring of the device to the native mitral annulus. Valve leaflets are made of bovine pericardium. The Cardiovalve implant has a very low left ventricle (LV) protrusion footprint thus reducing the risk of LV outflow tract obstruction and/or interference with the LV. The Cardiovalve delivery system (DS) is designed for transfemoral delivery of the Implant with transseptal access to the left atrium. The catheter assembly is used to center the implant relative to the native mitral valve plane and align it with the left ventricual apex-to-base axis. After valve implantation, the delivery system is withdrawn.

ELIGIBILITY:
General Inclusion Criteria

1. Age ≥ 18 years
2. NYHA functional II, III or ambulatory IV
3. Severe mitral regurgitation (MR grade 3-4+)
4. Subject is on optimal guideline-directed medical therapy for heart failure for at least 30 days or CRT if indicated.
5. Elevated risk for conventional open mitral valve repair or replacement surgery in the consideration of the site Heart Team (including a cardiac surgeon, a cardiologist and imaging specialist as a minimum) based on STS/Euro Score II (per MVARC Part 1), frailty and co-morbidities.
6. Able to undergo Transesophageal Echocardiography (TEE).
7. Subject understands the study requirements and the treatment procedures and provides written Informed Consent before any study-specific tests or procedures are performed.
8. The subject commits to return for the scheduled post-operative follow-up visits at the hospital.

   Anatomical Inclusion Criteria
9. Suitable for femoral access procedure and trans septal catheterization
10. Native mitral valve geometry and size and LV outflow tract characteristics compatible with the Cardiovalve (as assessed by the independent Screening Committee)

Cardiovascular Exclusion Criteria

1. Prior stroke or TIA within 3 months or Modified Rankin Scale ≥4 disability
2. Acute myocardial infarction within the previous 30 days
3. Any prior heart valve surgery or transcatheter mitral intervention
4. Any percutaneous cardiovascular intervention, cardiovascular surgery, or carotid surgery within 30 days
5. Rheumatic heart disease or endocarditis within the previous 3 months
6. Hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, or any other structural heart disease causing heart failure other than dilated cardiomyopathy of either ischemic or non-ischemic etiology
7. Existence of inferior vena cava filter or atrial septal device (contraindicating femoral access and transseptal catheterization)
8. Untreated clinically significant coronary artery disease requiring revascularization
9. Tricuspid valve disease requiring surgery or severe tricuspid regurgitation
10. Aortic or pulmonic valve disease requiring surgery
11. CRT/ICD implant within 30 days

    Anatomical Exclusion Criteria (assessed by pre-procedural imaging)
12. Left Ventricular Ejection Fraction (LVEF) <30%
13. LV end diastolic diameter > 70mm
14. Significant abnormalities of the mitral valve and sub-valvular apparatus.
15. Severe mitral annular or leaflets calcification
16. Left atrial or LV thrombus or vegetation
17. Severe right ventricular dysfunction
18. Severe tricuspid or aortic valve disease

    General Exclusion Criteria
19. Subject who is currently participating in an investigational study, other than this study
20. Hemodynamic instability defined as systolic pressure < 90mmHg or the need for inotropic support or intra-aortic balloon pump or other hemodynamic support device, or any mechanical heart assistance
21. Subject has contrast agent hypersensitivity that cannot be adequately pre-medicated, has an allergy to Nitinol alloys (nickel and titanium), or has intolerance to antiplatelet, anticoagulant, or thrombolytic medications
22. Bleeding diathesis or hypercoagulable state
23. Active peptic ulcer or active gastrointestinal bleeding
24. Pulmonary artery systolic pressure >70 mmHg
25. Patients with renal insufficiency (creatinine > 2.5 mg/dL)
26. Need for emergent or urgent surgery for any reason or any planned cardiac Surgery within the next 12 months
27. Subject with hepatic insufficiency
28. Subject has a co-morbid illness that may result in a life expectancy of less than one year
29. Active infection that requires antibiotic therapy
30. Subject is pregnant, breastfeeding or intend to become pregnant within one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-04-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary safety endpoint is freedom from all-cause mortality and major adverse events | 30 days, 3 Months, 6 Months, 12 Months, and 24 Months
  Freedom from all-cause mortality, all cause hospitalization, major adverse cardiac events (MACE), major device- or procedure- related serious adverse events

SECONDARY OUTCOMES:
Technical success | Intraoperative, 30 Days
  Technical success:
  I. Absence of procedural mortality
  II. Delivery and deployment of the device in the correct position and retrieval of delivery catheter, without significant mitral stenosis, LVOT obstruction or paravalvular MR documented by intraoperative imaging [Time Frame:Intraoperative]
  III. Freedom from emergency surgery or reintervention related to the device or access procedure [Time Frame: 30 days]
Device Success | Intraoperative
  I. Absence of procedural mortality or stroke
  II. Proper placement and positioning of the device
  III. Freedom from unplanned surgical or interventional procedures related to the device or access procedure
Device Success | 30 days, 3 Months, 6 Months, 12 Months, and 24 Months
  IV. Continued intended safety and performance of the device including:
  1. No evidence of structural or functional failure
  2. No specific device-related technical failure issues and complications
  3. Reduction in MR grade to either optimal (0+ to trace) or acceptable (reduced by at least 1 grade from baseline with no more than 2+ MR). Number of patients with reduction in MR grade from baseline
Patient Success | 30 days, 3 Months, 6 Months, 12 Months, and 24 Months
  I. Device success (either optimal or acceptable) II. Patient returned to the pre-procedural setting
  * III. Freedom from rehospitalizations or reinterventions for the underlying condition (e.g., mitral regurgitation, worsening of heart failure)
  * IV. Improvement from baseline in NYHA functional class Number of patients with improvement in NYHA class
  * V. Six minute walk test Increase in distance (m) from baseline
  * VI. Improvement from baseline in quality-of-life (Kansas City Cardiomyopathy Questionnaire improvement by ≥ 10)

CONTACTS AND LOCATIONS:
Overall Officials: Georg Nickenig, Principal Investigator — Bonn Clinic
Locations (11):
- Germany (5):
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Herzzentrum der Uniklinik Köln, Cologne
  - Studienzentrale der Medizinische Klinik II Universitäres Herzzentrum Lübeck, Lübeck
  - Universitaet_Mainz, Mainz
  - Klinikum der Universität München LMU, München
- Hygea, Athens, Greece
- Italy (5):
  - Maria Cecilia Hospital, Cotignola
  - Fondazione Toscana G. Monasterio-Ospedale del Cuore, Massa
  - San Raffaele Hospital, Milan
  - Policlinico San Donato, Milan
  - A.O.U. Pisana, Pisa

IPD SHARING:
Plan to Share IPD: No